CLINICAL TRIAL: NCT03739372
Title: A Pilot Trial Testing the Clinical Benefit of Using Molecular Profiling to Determine an Individualized Treatment Plan in Children and Young Adults With High Grade Glioma (Excluding Diffuse Intrinsic Pontine Glioma)
Brief Title: Clinical Benefit of Using Molecular Profiling to Determine an Individualized Treatment Plan for Patients With High Grade Glioma
Acronym: PNOC008
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Pacific Pediatric Neuro-Oncology Consortium (Other); The V Foundation for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 170827; PNOC008 (Other: Pacific Pediatric Neuro-Oncology Consortium (PNOC))
Record Dates: First submitted 2018-11-02; First posted 2018-11-13 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Glioma; Glioma of Brain; Cancer; Pediatric Cancer; Pediatric Brain Tumor; Astrocytoma; Glioblastoma; Hemispheric
Keywords: High-grade glioma; whole exome sequencing; WES; genomics; RNA sequencing
MeSH Terms: conditions — Glioma; Neoplasms; Astrocytoma; Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Newly diagnosed HGG (Stratum A) (Experimental): Children and young adults with newly diagnosed HGG receive an individualized treatment plan. Each treatment is different and depends on what the Specialized Tumor Board recommends depending on the molecular profile of the patient's tumor.
  Interventions: Other: Specialized tumor board recommendation
- Diffuse midline HGG (Stratum B) (Experimental): Children and young adults with diffuse midline high grade gliomas receive an individualized treatment plan. Each treatment is different and depends on what the Specialized Tumor Board recommends depending on the molecular profile of the patient's tumor.
  Interventions: Other: Specialized tumor board recommendation

INTERVENTIONS:
Other: Specialized tumor board recommendation — Based on the molecular profile, the specialized tumor board will determine an individualized treatment recommendation for each patient using up to four FDA approved drugs. In special circumstances, Investigational new drug (IND) study agents may be used.

SUMMARY:
This is a 2 strata pilot trial within the Pacific Pediatric Neuro-Oncology Consortium (PNOC).

The study will use a new treatment approach based on each patient's tumor gene expression, whole-exome sequencing (WES), targeted panel profile (UCSF 500 gene panel), and RNA-Seq. The current study will test the efficacy of such an approach in children with High-grade gliomas HGG.

DETAILED DESCRIPTION:
For children with High-grade gliomas (HGG) including HGG presenting within the midline structures of the brain and spine, outcome remains poor and the majority of children die from this disease. The current study will use a new treatment approach based on each patient's tumor gene expression, whole-exome sequencing (WES), targeted panel profile (UCSF 500 gene panel), and RNA-Seq. This treatment strategy has shown promising results in adult patients with solid tumors and is currently being explored in children with DIPG, neuroblastoma and other solid tumors. The current study will test the efficacy of such an approach in children with HGG for which outcomes remain dismal.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed HGG (including midline HGG but excluding DIPG), who undergo tissue collection as part of standard of care. HGG is defined as either World Health Organization (WHO) grade III or IV, or testing positive for H3K27M mutation. Patients with disseminated disease are not eligible, and MRI of the spine must be performed if disseminated disease is suspected by the treating physician. Primary spinal cord tumors are eligible.
* Enrollment within 3 weeks of the start of radiation therapy.
* Start of radiation therapy within 6 weeks from initial tissue diagnosis.
* Age ≤ 21 years
* Karnofsky score ≥ 50 for patients ≥ 16 years of age and Lansky score ≥ 50 for patients ≤15 years of age. Patients who are unable to walk because of paralysis but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Adequate tissue for molecular profiling (see Section 8 of the protocol for full details)
* The effects of the current treatment paradigm on the developing human fetus are unknown. For this reason, females of child-bearing potential and males must agree to use adequate contraception: hormonal or barrier method of birth control; abstinence prior to study entry and for the duration of study participation, and 30 days after completion of study drug administration. Should a female become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Males treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 30 days after completion of study drug administration.
* Adequate neurologic function defined as: Patients with seizure disorder may be enrolled if seizures are well controlled.
* Ability by patient or parent/legal guardian to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

* Patients who are currently enrolled on another therapeutic clinical trial. Individual cases should be discussed with the study chair.
* Patients who are currently taking any anti-cancer directed therapy. Steroids are not considered anti-cancer therapy. The use of temozolomide during radiation therapy is allowed at standard dosing (maximum 75 to 90 mg/m^2 daily for a total of 42 days). Any other schedule(s) need to be discussed with the study chair.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Female patients of childbearing potential must not be pregnant or breast-feeding. Female patients of childbearing potential must have a negative serum or urine pregnancy test prior to the start of therapy (as clinically indicated).
* Patients with inability to return for follow-up visits or obtain follow-up studies required to assess toxicity to therapy. Telemedicine visits are acceptable.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Estimated)
Dates: Start 2018-11-28 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
12 month Progression Free Survival (PFS) for Stratum A | Up to 12 months
  Progression Free Survival will be determined from date of confirmation of response to first evidence of progression or death at the 12 month time point.
12 month Overall Survival (OS) for Stratum B | Up to 12 months
  Overall survival will be determined from the date of histological diagnosis to time of death at the 12 month time point.

SECONDARY OUTCOMES:
Frequency of Adverse Events | From beginning of enrollment up to 30 days post end of treatment.
  Toxicity will be described by reporting Adverse Events (AE). Events will be assessed according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) v5.0. All study-related and unrelated AEs will be collected and reported, together with their maximum intensity among all recorded respective AE.
Frequency of Serious Adverse Events | From beginning of enrollment up to 30 days post end of treatment.
  Toxicity will be described by reporting Serious Adverse Events (SAE). Events will be assessed according to the NCI CTCAE v5.0. All study-related and unrelated Serious Adverse Events (SAE) will be collected and reported, together with their maximum intensity among all recorded respective SAE.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Mueller, MD, PhD, MAS, Principal Investigator — University of California, San Francisco
Locations (12):
- United States (12):
  - University of California, San Diego Rady Children's Hospital, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Children's Hospitals and Clinics of Minneapolis, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Children's Hospital Of Philadelphia, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data after de-identification.
Supporting Information: Study Protocol